CLINICAL TRIAL: NCT00069446
Title: An Exploratory, Double-Blind, Randomized, Placebo Controlled Study Evaluating Topical Recombinant Human Vascular Endothelial Growth Factor (Telbermin) for Induction of Healing of Chronic, Diabetic Foot Ulcers
Brief Title: A Study Evaluating Topical Recombinant Human Vascular Endothelial Growth Factor (Telbermin) for Induction of Healing of Chronic, Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: VGF2763g
Record Dates: First submitted 2003-09-25; First posted 2003-09-26 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Foot Ulcer
Keywords: Diabetes; Diabetic; Diabetic Foot Ulcer
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus; Diabetic Foot

INTERVENTIONS:
Drug: rhuMAb VEGF (telbermin)

SUMMARY:
This is a Phase I, double blind, randomized, placebo-controlled study that will enroll approximately 50 adult subjects with Type 1 or Type 2 diabetes mellitus and chronic, diabetic foot ulcers. The study will be conducted at approximately 12 investigational sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* 18-80 years old
* For females of childbearing potential, use of an effective method of contraception: abstinence; surgical sterilization; oral contraceptives; barrier contraception with either a condom, sponge, or diaphragm in conjunction with spermicidal gel; an intrauterine device (IUD); or contraceptive hormone implant or patch
* Type 1 or 2 diabetes mellitus
* Single, full-thickness (i.e., extending into the subcutaneous tissue or beyond) ulcer of the foot below the malleolus that does not involve bone, tendons, ligaments, or muscle
* Chronic ulcer with a duration of ≥ 4 weeks but < 6 months
* Ulcer area with sharp debridement of ≥ 1.0 cm^2 and ≤ 4.0 cm^2
* Ankle-brachial index (ABI) of ≥ 0.6 and ≤ 1.2 on the study foot
* Glycosylated hemoglobin A1c (HbA1c) of ≤ 12%

Exclusion Criteria:

* History of neoplasia or current neoplasia (with the exception of non-melanoma skin cancer)
* Proliferative diabetic retinopathy or wet age-related macular degeneration
* Active ulcer infection or cellulitis of any ulcer
* Ulcers with an etiology not related to diabetes (e.g., thermal, chemical, radiation insult)
* Connective tissue disease
* Active osteomyelitis of the study foot
* Subjects with ulcers related to an incompletely healed amputation wound
* Subjects with Charcot or other deformity of the study foot involving the study ulcer
* Immunosuppressive treatment, including radiation therapy, non-inhaled corticosteroids (inhaled corticosteroid ≤ 1000 ug daily dose is acceptable), and chemotherapy
* Pregnancy or lactation
* Multiple ulcers in the study foot
* Renal failure (serum creatinine of >3.0 mg/dL)
* Poor nutritional status (albumin of <3.0 g/dL)
* Known hypersensitivity to any ingredients of telbermin, placebo, or vehicle, including excipients in the formulation of telbermin or placebo gel (trehalose dihydrate, polysorbate 20, succinic acetic acid, succinic acetic acid disodium, and hexahydrate)
* Known prior inability to complete required study visits during treatment period
* Use of any other investigational drug or therapy on the study foot within the past month
* Previous use of a platelet-derived or other growth factors on the study ulcer within the past 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-08 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant hypotension.

SECONDARY OUTCOMES:
Incidence of clinically significant ulcer infection defined by increased discharge and malodorous exudates from the ulcer, fever, and a white blood cell (WBC) count of >10,000/uL
Development of anti telbermin antibodies
Incidence of adverse events
Percent reduction in total ulcer surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Breen, Ph.D., Study Director — Genentech, Inc.